CLINICAL TRIAL: NCT00846378
Title: The Mechanism of Ischemic Post-conditioning in Humans: Minimizing Reperfusion Injury in Patients With Acute Myocardial Infarction
Brief Title: Minimizing Reperfusion Injury in Patients With Acute Myocardial Infarction
Acronym: PCinAMI
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended for potential change in protocol to include different imaging modalities
Sponsor: University of Cincinnati (Other)
Collaborators: Cardiology Research UBC (Other)
Responsible Party: Principal Investigator, Tarek Helmy, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCIRB07051803
Record Dates: First submitted 2008-04-16; First posted 2009-02-18 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Acute Myocardial Infarction
Keywords: ST segment elevation myocardial infarction (STEMI); timed balloon inflations; post conditioning
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post conditioning (Experimental): After 30 seconds of re-established coronary flow following the therapeutic balloon dilatation and deflation, the same balloon will be re-inflated for 30 seconds and then again deflated for 30 seconds. The balloon should be inflated to only occlude the coronary artery. This procedure of balloon inflation/deflation will be performed a total of 3 to 4 times.
  Interventions: Procedure: Post conditioning
- Usual Care (Active Comparator): Usual care for treatment of thrombolysis in myocardial infarction (TIMI) 0 to TIMI 1 flow in occluded infarct related artery. Usual care includes reperfusion of the artery per operator discretion, i.e. primary stenting, thrombectomy, balloon inflation/deflation without timed intervals.
  Interventions: Procedure: Usual Care for STEMI

INTERVENTIONS:
Procedure: Post conditioning — after 30 seconds of re-established coronary flow following the therapeutic balloon dilatation and deflation, the same balloon will be re-inflated for 30 seconds and then again deflated for 30 seconds. This procedure of balloon inflation/deflation will be performed a total of 3 to 4 times.
  Arms: Post conditioning
Procedure: Usual Care for STEMI — Usual care for treatment of TIMI 0 to TIMI 1 flow in occluded infarct related artery. Usual care includes reperfusion of the artery per operator discretion, i.e. primary stenting, thrombectomy, balloon inflation/deflation without timed intervals.
  Arms: Usual Care

SUMMARY:
The size of a heart attack will be decreased by the use of timed balloon inflations to open the blocked blood vessel.

DETAILED DESCRIPTION:
The intervention of "post conditioning" at the time of reperfusion, in patients with acute myocardial infarction (AMI), will attenuate the degree of ischemia-reperfusion injury, as manifested by infarct size. This intervention is hypothesized to be safe in humans.

ELIGIBILITY:
Inclusion Criteria:

* STEMI
* Onset of symptoms within 6 hours
* TIMI 0 to TIMI 1 flow in infarct related artery

Exclusion Criteria:

* collaterals to infarct related artery
* previous infarct in related territory
* thrombolytics
* cardiogenic shock
* TIMI 2 to TIMI 3 flow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Quantitation of infarct size will be done using a modification of University Hospital's standard Single-photon emission computed tomography (SPECT) quantitation software | 6 weeks
Echocardiograms will be analyzed to evaluate left ventricular function. Standard techniques will be used to quantitate ejection fraction and the percentage of left ventricular circumference that is hypokinetic or dyskinetic. | 6 weeks
Venous blood samples troponin, creatine phosphokinase (CPK). This will be done to follow enzyme release and washout, and area data will be available and infarct size/risk area ratios in control and post-conditioning subjects will be compared. | baseline, every 8 hours x 3
ECG ST segment resolution immediate post percutaneous coronary intervention(PCI), and daily x 3. | baseline, up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Helmy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States